CLINICAL TRIAL: NCT06327555
Title: Comparison of the Efficacy of Telerehabilitation and In-person Rehabilitation Based on Wearable Devices After ACLR Surgery: a Multicenter Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking Union Medical College Hospital (Other); Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2023132
Record Dates: First submitted 2024-03-17; First posted 2024-03-25 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2024-09

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: ACLR; Telerehabilitation
MeSH Terms: interventions — Telerehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- in-person rehabilitation group (Other): The in-person rehabilitation group takes a face-to-face approach, with therapists providing outpatient rehabilitation instruction twice a week for six weeks.
  Interventions: Other: in-person rehabilitation
- telerehabilitation group (Experimental): The telerehabilitation group uses software and sensors to provide remote postoperative rehabilitation guidance.
  Interventions: Other: telerehabilitation

INTERVENTIONS:
Other: telerehabilitation — The telerehabilitation group uses smart wearables and mobile apps worn around the knee joint to perform telerehabilitation at home. Both sets of training sessions are identical.
  Arms: telerehabilitation group
Other: in-person rehabilitation — The in-person rehabilitation group uses a face-to-face approach, with therapists providing outpatient rehabilitation guidance to patients three times a week for six weeks. After that, patients exercise at home according to the rehabilitation manual.
  Arms: in-person rehabilitation group

SUMMARY:
Purpose: Investigate whether telerehabilitation based on wearable devices is clinically as effective as in-person rehabilitation for ACLR patients.

Subjects: 164 patients aged ≥18 years who underwent ACLR. Design: A mixed-block randomization method was used to randomly assign participants to two groups: the telerehabilitation group and the in-person rehabilitation group, with a 50% probability of assignment to each group. All participants received standard postoperative rehabilitation training with identical content. The telerehabilitation group received postoperative telerehabilitation guidance via software and sensors. The in-person rehabilitation group received therapist-administered treatment with three rehabilitation sessions per week. All participants underwent regular follow-ups (1 day preoperatively, 3 months postoperatively, and 6 months postoperatively).

Primary outcome measure: The primary outcome measure was the Lysholm score. Secondary outcome measures included the IKDC score, Tegner Activity Scale, SF-36 questionnaire, VAS score, and isokinetic muscle strength of the knee joint.

DETAILED DESCRIPTION:
Purpose: Investigate whether telerehabilitation based on wearable devices is clinically as effective as in-person rehabilitation for ACLR patients.

Subjects: Participants: This study recruited 164 participants (aged ≥18 years) undergoing ACLRsurgery;

Inclusion criteria:

(1) Age range 18-60 years; (2) First-time unilateral ACLR surgery or ACLR combined with meniscus resection surgery; (3) No other lower limb joint injuries at the same time; (4) Possession of an internet-connected mobile device capable of using a mobile application; (5) Alert and oriented, with no communication impairments; Exclusion Criteria: (1) Patients undergoing revision surgery; (2) Patients who have previously undergone other lower limb surgeries; (3) Patients scheduled for another lower limb surgery within the next 6 months; (4) Patients with concomitant knee ligament injuries or severe structural damage beyond meniscal tears; (5) Patients with other comorbidities that may interfere with rehabilitation exercises; (6) Patients undergoing acute-phase surgery; (7)Patients undergoing acute surgery.

Protocol: Participants were randomly assigned to two groups using a mixed-block randomization method: the telerehabilitation group and the in-person rehabilitation group. The allocation probability for both groups was 50%. All participants received routine outpatient diagnosis and treatment. Postoperative rehabilitation training used a standardized postoperative rehabilitation training protocol with identical content. The telerehabilitation group received postoperative telerehabilitation guidance via software and sensors. The in-person rehabilitation group received three face-to-face rehabilitation sessions per week. All participants underwent regular follow-ups (1 day preoperatively, 3 months postoperatively, and 6 months postoperatively).

Primary outcome measure: The primary outcome measure was the Lysholm score. Secondary outcome measures included the IKDC score, Tegner Activity Scale, SF-36 questionnaire, VAS score, isokinetic muscle strength of the knee joint, and muscle strength symmetry.

ELIGIBILITY:
Inclusion Criteria:

(1) Age range 18-60 years; (2) First-time unilateral ACLR surgery or ACLR combined with meniscus resection surgery; (3) No other lower limb joint injuries at the same time; (4) Possession of an internet-connected mobile device capable of using a mobile application; (5) Alert and oriented, with no communication impairments;

Exclusion Criteria:

(1) Patients undergoing revision surgery; (2) Patients who have previously undergone other lower limb surgeries; (3) Patients scheduled for another lower limb surgery within the next 6 months; (4) Patients with concomitant knee ligament injuries or severe structural damage beyond meniscal tears; (5) Patients with other comorbidities that may interfere with rehabilitation exercises; (6) Patients undergoing acute-phase surgery; (7)Patients undergoing acute surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Lysholm score | From before ACLR surgery to 6 months post-surgery.
  Used to assess knee joint function, with a score range of 0-100, where a higher score indicates better knee joint function.

SECONDARY OUTCOMES:
IKDC score | From before ACLR surgery to 6 months post-surgery.
  Used to assess knee joint function, with a score range of 0-100. The higher the score, the better the knee joint function.
Tegner score | From before ACLR surgery to 6 months post-surgery.
  Used to assess motor function. The range is 0-10, with higher scores indicating better knee function.
VAS score | From before ACLR surgery to 6 months after surgery.
  Used to assess pain levels. The range is 0-10, with higher scores indicating higher pain levels.
Short Form-36 Health Survey(SF-36) | From before ACLR surgery to 6 months post-surgery.
  Used to assess quality of life. There are 9 subscales, each with a score range of 0-100, with higher scores indicating better knee function.
Peak torque and symmetry of knee flexors and extensors | From before ACLR surgery to 6 months after surgery.
  Used to assess knee muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: quan J Wang, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- quan Jian Wang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No